CLINICAL TRIAL: NCT00399386
Title: ECG Recordings From EP Study, Defibrillator Implantation or Ablation Procedure in Paediatric Population
Brief Title: Electrocardiogram (ECG) Recordings in Paediatric Population
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: DN-05039
Record Dates: First submitted 2006-11-10; First posted 2006-11-14 (Estimated); Last update posted 2017-02-16 (Actual); Status verified 2009-10

CONDITIONS: Arrhythmia
Keywords: S ICD; ICD; Ablation; EP study; Paediatric; ECG
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Procedure: EP
Procedure: ICD
Procedure: Ablation

SUMMARY:
The primary goal of this protocol is to collect ECG signals from paediatric patients using 4 surface electrodes placed in the configurations proposed for the Cameron Health, Inc. subcutaneous implantable defibrillator (S-ICD) system. These signals will then be used to test the S-ICD system for future use in paediatric patients.

DETAILED DESCRIPTION:
The surface ECGs collected from pediatric patients in normal sinus rhythm and a variety of ventricular and atrial arrhythmias will be used as test signals for the development of the S-ICD system. These signals will be collected from patients undergoing electrophysiology (EP) study, transvenous defibrillator implantation or ablation procedures

ELIGIBILITY:
Inclusion Criteria:

* Patients < 18 years of age
* Patient scheduled for an EP study, implantation of an ICD or for an ablation procedure

Exclusion Criteria:

* Patients whose parents/guardians do not sign an informed consent

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients at the Bristol Royal Hospital for Children
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2006-11; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Graham Stuart, MD, Principal Investigator — Bristol Childrens' Hospital
Locations (1):
- Bristol Childrens' Hospital, Bristol, Avon, United Kingdom